CLINICAL TRIAL: NCT00001962
Title: A Pilot Study of Recombinant Humanized Anti-Interleukin (IL-2) Receptor Antibody (Daclizumab) in Patients With Moderate Aplastic Anemia, Pure Red Cell Aplasia, or Diamond Blackfan Anemia
Brief Title: A Study to Determine Whether Therapy With Daclizumab Will Benefit Patients With Bone Marrow Failure
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: DSMB recommended closing the study and publishing the results
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 000029; 00-H-0029 (Other: NIH NHLBI)
Record Dates: First submitted 2000-01-18; First posted 2000-01-19 (Estimated); Results first posted 2015-05-14 (Estimated); Last update posted 2021-07-09 (Actual); Status verified 2015-04

CONDITIONS: Aplastic Anemia; Pure Red Cell Aplasia; Diamond Blackfan Anemia
Keywords: Immunosuppression; T-cells; Hematopoiesis; Monoclonal Antibody Therapy; Immunosuppressive Therapy; Aplastic Anemia
MeSH Terms: conditions — Anemia, Aplastic; Red-Cell Aplasia, Pure; Anemia, Diamond-Blackfan | interventions — Daclizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Daclizumab in participants with a bone marrow failure syndrome (Experimental): daclizumab, 1 mg/kg, will be given for a total of 5 intravenous infusions. These subjects may be diagnosed with moderate aplastic anemia, pure red cell aplasia, Diamond Blackfan anemia, relapse and refractory severe aplastic anemia will receive treatment. The subjects will be seen and receive the daclizumab infusion biweekly during the treatment period.
  Interventions: Drug: Daclizumab

INTERVENTIONS:
Drug: Daclizumab — Daclizumab, 1mg/kg, every 2 weeks for a total of 5 infusions.
  Other Names: Zenapax

SUMMARY:
Participants in this study are suffering from rare and serious blood disorders. In aplastic anemia, the bone marrow stops producing red blood cells, platelets, and white blood cells. In pure red cell aplasia, the bone marrow stops producing red cells, and in amegakaryocytic thrombocytopenic purpura, the bone marrow stops producing platelets.

Current treatment approaches for these disorders include bone marrow transplant and/or immunosuppression. However, bone marrow transplant is not always possible, and immunosuppression has serious side effects.

This study will investigate whether daclizumab can be used to treat these disorders. Daclizumab is a genetically engineered human antibody that blocks the interleukin-2 receptor on immune cells. It has been used successfully in many transplant patients to reduce the rate of organ rejection.

Participants will undergo a complete history and physical examination. A bone marrow aspiration and biopsy will be performed to confirm the type of bone marrow failure. About 5 tablespoons of blood will be drawn for baseline tests and research purposes. Daclizumab will be administered every 2 weeks by vein in a 30-minute infusion. The first dose will be given at NIH and the next four may be given at NIH or by the participant's primary hematologist. The treatment will last 8 weeks. Participants must also see their referring physician or NIH physicians every 2 weeks for blood counts. In the fourth and eighth weeks of the study and at the 3-month follow-up visit, 2 tablespoons of blood will be drawn at NIH. At the 1-month follow-up visit to NIH, 5 tablespoons of blood will be drawn and another bone marrow aspiration and biopsy performed.

Risks from bone marrow aspiration and biopsy and blood draws include discomfort. Daclizumab is usually well-tolerated; however, it may weaken immunity against certain bacteria and viruses.

DETAILED DESCRIPTION:
Many bone marrow failure syndromes in humans are now recognized to result from immunological mechanisms. These diseases include aplastic anemia; single hematopoietic lineage failures such as pure red cell aplasia, Diamond Blackfan Anemia, agranulocytosis, and amegakaryocytic thrombocytopenic purpura; and some types of myelodysplasia. Patients with these conditions, who may suffer variable degrees of anemia, leukocytopenia, and thrombocytopenia, alone or combination, have been shown to respond to a wide variety of immunosuppressive agents, ranging from corticosteroids to cyclosporine (CSA) and antithymocyte globulin (ATG). However, except for severe aplastic anemia, which has been shown to be appropriately treated with either bone marrow transplantation or a combination of ATG and CSA, single agents or regimens have usually not been applied systematically to other immune-mediated hematologic diseases. In an effort to discover other and especially less toxic treatments for immunologically-mediated bone marrow diseases, we seek to apply a new therapy, a humanized anti-interleukin-2 receptor (lL-2R) monoclonal antibody (mAb ), to a subset of patients with bone marrow failure. Anti-IL-2R mAb acts against activated lymphocytes, thus sharing an important mechanism of action with ATG. However, the mAb is much less toxic than ATG and may be administered to outpatients at relatively infrequent intervals (every 2 weeks).

The primary objective is to test the efficacy of anti-IL-2R mAb (daclizumab), we propose to treat four groups of patients: 1) moderate aplastic anemia, 2) single lineage failure states including pure red cell aplasia or Diamond Blackfan anemia, 3) relapse of severe aplastic anemia and 4) refractory severe aplastic anemia not responding to both horse and rabbit ATG/CsA. Subjects will receive daclizumab once every other week for a total of 5 doses. Patients relapsing after response to initial treatment may be treated with 2 additional courses of daclizumab. In November 2005, the relapsed and refractory severe aplastic anemia arms were closed by the Data and Safety Monitoring Board (DSMB) for lack of efficacy. In October 2008, the moderate aplastic anemia arm was closed by the DSMB when the data was determined sufficient for making statistical inferences regarding the original hypotheses. In October 2008, accrual to the Diamond Blackfan anemia arm was closed by the DSMB for lack of accrual.

The Primary endpoint is hematologic response at 3 months. Secondary endpoints include transfusion dependence, overall survival, life threatening toxicity, transformation-free survival, and response duration.

ELIGIBILITY:
-INCLUSION CRITERIA:

1. Acquired pure red cell aplasia requiring red blood cell (RBC) transfusions defined by

   * anemia,
   * reticulocytopenia (reticulocyte count less than or equal to 50,000/mm(3))
   * and absent or decreased marrow erythroid precursors

   Acquired aplastic anemia of moderate severity (In October 2008, this arm was closed by the DSMB when the data was determined sufficient for making statistical inferences regarding the original hypotheses.

   Diamond Blackfan Anemia (DBA) (In October 2008, accrual of DBAs was closed by the DSMB for lack of accrual)

   Relapsed patients with severe aplastic anemia (In November 2005 this arm was closed by the DSMB for lack of efficacy)

   Refractory disease not responding to both horse and rabbit ATG/CsA (In November 2005 this arm was closed for lack of efficacy)
2. Age greater than or equal to 2 years old
3. Weight greater than 12 kg
4. Patients or their parent(s)/responsible guardian(s) must be able to comprehend and be willing to sign an informed consent.

EXCLUSION CRITERIA:

Current diagnosis or past history of myelodysplastic syndrome or Fanconi's anemia.

Known allergy to E.coli-derived products.

Persistent B19 parvovirus infection.

Evidence of uncontrolled infection.

Chronic or current clinically significant infection, including HIV positivity or hepatitis B and C virus infection.

Significant other diseases, congestive heart failure (greater than New York Class II), poorly controlled diabetes mellitus, uncontrolled cardiac arrhythmias.

Subjects with cancer who are on active chemotherapeutic treatment or who take drugs with hematological effects will not be eligible

A moribund status or concurrent hepatic, renal, cardiac, metabolic disease of such severity that death within 1-4 weeks from initiation of therapy is likely.

Recent major surgery.

Treatment with an investigational agent other than hematopoietic growth factors within 4 weeks of study entry.

Psychiatric, affective, or other disorder that may compromise the ability to give informed consent or to cooperate in a research study.

Pregnancy or lactation.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 1999-11; Primary Completion 2009-08 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neal Young, MD, Principal Investigator — NIH National Heart, Lung, and Blood Institute
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Young NS, Barrett AJ. The treatment of severe acquired aplastic anemia. Blood. 1995 Jun 15;85(12):3367-77. No abstract available. PMID 7780125
- [Background] Young NS, Maciejewski J. The pathophysiology of acquired aplastic anemia. N Engl J Med. 1997 May 8;336(19):1365-72. doi: 10.1056/NEJM199705083361906. No abstract available. PMID 9134878
- [Background] Maciejewski JP, Hibbs JR, Anderson S, Katevas P, Young NS. Bone marrow and peripheral blood lymphocyte phenotype in patients with bone marrow failure. Exp Hematol. 1994 Oct;22(11):1102-10. PMID 7925777
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/detail/B_2000-H-0029.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Daclizumab in Bone Marrow Failure Syndromes: Daclizumab, 1 mg/kg, will be given for a total of 5 intravenous infusions in participants with a bone marrow failure syndrome. These subjects may be diagnosed with moderate aplastic anemia, pure red cell aplasia, Diamond Blackfan anemia, relapse and refractory severe aplastic anemia will receive treatment. The subjects will be seen and receive the daclizumab infusion biweekly during the treatment period.
Period: Overall Study
Arm/Group | Daclizumab in Bone Marrow Failure Syndromes
Started | 100
Completed | 72
Not Completed | 28
Not completed — Lack of Efficacy | 18
Not completed — Lack of Accrual | 6
Not completed — Death | 1
Not completed — Lost to Follow-up | 2
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Daclizumab in Bone Marrow Failure Syndromes
Number analyzed (Participants) | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 27
  Between 18 and 65 years | 57
  >=65 years | 16
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49
  Male | 51

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Hematologic Response Following Daclizumab in Patients With Moderate Aplastic Anemia (MAA) and Pure Red Cell Aplasia (PRCA).
Description: Number of participants with hematologic response at 3 months following Daclizumab, 1 mg/kg, will be given for a total of 5 intravenous infusions to subjects diagnosed with moderate aplastic anemia (MAA), pure red cell aplasia (PRCA), Diamond Blackfan anemia (DBA), relapse and refractory severe aplastic anemia (SAA) will receive treatment.
  A complete hematologic response will be considered an achievement of normal blood counts. A partial response was defined as any response less than a complete response. The primary endpoint was a hematologic response in at least one affected peripheral blood count parameter, as determined by 3 separate measurements in the first 12 weeks after completion of the infusion.
Time Frame: 3 months
Population: The daclizumab hematologic response was evaluated for subjects diagnosed with moderate aplastic anemia (MAA) and pure red cell aplasia (PRCA). The Diamond Blackfan arm was closed due to lack of accrual. Relapse and Refractory Severe Aplastic Anemia (SAA) was closed to lack of efficacy.
Measure: Number; unit: participants
Groups:
- Daclizumab in Participants With a Bone Marrow Failure Syndrome: Daclizumab, 1 mg/kg, will be given for a total of 5 intravenous infusions in participants with a bone marrow failure syndrome. These subjects may be diagnosed with moderate aplastic anemia, pure red cell aplasia, Diamond Blackfan anemia, relapse and refractory severe aplastic anemia will receive treatment. The subjects will be seen and receive the daclizumab infusion biweekly during the treatment period.
Arm/Group | Daclizumab in Participants With a Bone Marrow Failure Syndrome
Number analyzed (Participants) | 72
participants
  MAA Complete response | 6
  MAA Partial response | 13
  MAA No response | 26
  PRCA Complete response | 6
  PRCA Partial response | 4
  PRCA No response | 17

2. Secondary Outcome: Number of Participants That no Longer Required Blood Transfusion
Description: Number of participants that no longer required blood transfusion after receiving Daclizumab, 1 mg/kg, for a total of 5 intravenous infusions to subjects diagnosed with moderate aplastic anemia (MAA), pure red cell aplasia (PRCA), Diamond Blackfan anemia (DBA), relapse and refractory severe aplastic anemia (SAA) will receive treatment.
Time Frame: 5 years
Population: This was evaluated for subjects diagnosed with moderate aplastic anemia (MAA) and pure red cell aplasia (PRCA). The Diamond Blackfan anemia arm was closed due to the lack of accrual. The Relapse and Refractory Severe Aplastic Anemia (SAA) was closed due to lack of efficacy.
Measure: Number; unit: participants
Arm/Group | Daclizumab in Participants With a Bone Marrow Failure Syndrome
Number analyzed (Participants) | 72
participants
  MAA | 7
  PRCA | 28

3. Secondary Outcome: Overall Survival
Description: Overall Survival at end of study after receiving Daclizumab, 1 mg/kg, for a total of 5 intravenous infusions to subjects diagnosed with moderate aplastic anemia (MAA), pure red cell aplasia (PRCA), Diamond Blackfan anemia (DBA), relapse and refractory severe aplastic anemia (SAA) will receive treatment.
Time Frame: 5 years
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Daclizumab in Participants With a Bone Marrow Failure Syndrome
Number analyzed (Participants) | 72
Participants
  Deaths | 7
  Alive | 65

ADVERSE EVENTS:
Time Frame: 5 years
Arm/Group | Daclizumab in Participants With a Bone Marrow Failure Syndrome
All-Cause Mortality (participants affected / at risk) | 7/100
Serious Adverse Events (participants affected / at risk) | 9/100
Other Adverse Events (participants affected / at risk) | 40/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Daclizumab in Participants With a Bone Marrow Failure Syndrome (N=100)
infection (Immune system disorders) | 2 (2)
renal failure (Renal and urinary disorders) | 1 (1)
hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — Herpes zoster
elevated liver function tests (Hepatobiliary disorders) | 1 (1)
polycythemia (Blood and lymphatic system disorders) | 1 (1)
angina (Cardiac disorders) | 1 (1)
sinusitis (Infections and infestations) | 1 (1)
gastroenteritis (Infections and infestations) | 1 (1) — wound- infectious
myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Daclizumab in Participants With a Bone Marrow Failure Syndrome (N=100)
shortness of breath (Infections and infestations) | 9 (9)
headache (General disorders) | 11 (12)
diarrhea (Gastrointestinal disorders) | 7 (7)
pain (Musculoskeletal and connective tissue disorders) | 6 (6)
dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
edema (Cardiac disorders) | 14 (14) — periorbital, lower extremity
fatigue (General disorders) | 5 (5)
fever (General disorders) | 4 (4)
eczema (Skin and subcutaneous tissue disorders) | 1 (1)
blurred vision (Eye disorders) | 3 (3)
alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
rash (Skin and subcutaneous tissue disorders) | 14 (15)
pallor (General disorders) | 4 (4)
abdominal pain (Gastrointestinal disorders) | 2 (2)
gynecomastia (Endocrine disorders) | 1 (1)
nausea (Gastrointestinal disorders) | 11 (11)
mouth sores (Gastrointestinal disorders) | 7 (7)
gum bleeding (Blood and lymphatic system disorders) | 9 (9)
back pain (General disorders) | 6 (6)
tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1)
lightheadness (Nervous system disorders) | 4 (4)
depression (Nervous system disorders) | 1 (1)
knee pain (General disorders) | 3 (3)
upper respiratory tract infection (Infections and infestations) | 40 (48)
urinary tract infection (Infections and infestations) | 6 (6)
hepatic pain (General disorders) | 3 (3)
arthritis (Musculoskeletal and connective tissue disorders) | 2 (2)
cough (Respiratory, thoracic and mediastinal disorders) | 2 (4)
viral infection (Infections and infestations) | 1 (1) — localized earache
myalgia (General disorders) | 6 (6)
constipation (Gastrointestinal disorders) | 5 (5)
palpitations (Cardiac disorders) | 2 (2)
dizziness (General disorders) | 3 (3)
weight gain (General disorders) | 3 (3)
sclerodactyly (Skin and subcutaneous tissue disorders) | 1 (1)
hyperparathyroid (Endocrine disorders) | 1 (1)
petechiae (Blood and lymphatic system disorders) | 13 (13)
cramps (Musculoskeletal and connective tissue disorders) | 4 (4)
decreased potassium (Metabolism and nutrition disorders) | 1 (1)
hearing loss (Ear and labyrinth disorders) | 1 (1)
elevated hemoglobin (Blood and lymphatic system disorders) | 2 (2)
hemolysis (Blood and lymphatic system disorders) | 1 (1)
lower extremity edema (Cardiac disorders) | 1 (1)
peripheral vascular disease (Cardiac disorders) | 1 (1)
rosacea (Skin and subcutaneous tissue disorders) | 1 (1)
earache (Ear and labyrinth disorders) | 2 (2)
allergic reaction (Immune system disorders) | 7 (7)
elevated liver function tests (Hepatobiliary disorders) | 3 (3)
strept throat (Infections and infestations) | 1 (2)
post nasal drip (Immune system disorders) | 1 (1)
diaphoresis (General disorders) | 1 (1)
acne (Skin and subcutaneous tissue disorders) | 1 (1)
furuncle (Skin and subcutaneous tissue disorders) | 1 (1)
nail changes (Skin and subcutaneous tissue disorders) | 1 (1)
skin lesions (Skin and subcutaneous tissue disorders) | 3 (3)
hypothyroidism (Endocrine disorders) | 1 (1)
anorexia (Gastrointestinal disorders) | 1 (1)
esophageal stricture (Gastrointestinal disorders) | 1 (1) — Barretts esophageal stricture
abdominal discomfort (Gastrointestinal disorders) | 3 (3)
duodenal ulcer (Gastrointestinal disorders) | 1 (1)
gingival hyperplasia (Gastrointestinal disorders) | 1 (1)
heartburn (Gastrointestinal disorders) | 1 (1)
endometrial benign polyp (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
ear bleeding (Blood and lymphatic system disorders) | 1 (1)
trauma bleeding (Blood and lymphatic system disorders) | 1 (1)
vaginal bleeding (Blood and lymphatic system disorders) | 2 (2)
blood blisters (Blood and lymphatic system disorders) | 1 (1)
blood in stool (Blood and lymphatic system disorders) | 3 (3)
bruising (Blood and lymphatic system disorders) | 9 (9)
epistaxis (Blood and lymphatic system disorders) | 6 (6)
heavy menses (Blood and lymphatic system disorders) | 2 (2)
retinal hemorrhage (Blood and lymphatic system disorders) | 1 (1)
subconjunctival hemorrhage (Blood and lymphatic system disorders) | 1 (1)
catheter related sepsis (Infections and infestations) | 1 (2)
gastritis (Infections and infestations) | 1 (1)
localized infection (Infections and infestations) | 4 (4)
strep throat (Infections and infestations) | 1 (2)
prostate malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
localized infection (Infections and infestations) | 1 (1) — swollen lymph nodes
neck stiffness (Musculoskeletal and connective tissue disorders) | 1 (1)
anxiety (Nervous system disorders) | 1 (1)
insomnia (Nervous system disorders) | 2 (2)
sensory neuropathy (Nervous system disorders) | 1 (1)
vertigo (Nervous system disorders) | 1 (1)
bone pain (General disorders) | 4 (4)
joint pain (General disorders) | 1 (2) — arthralgia
leg pain (General disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes